CLINICAL TRIAL: NCT00437580
Title: Impact of Probiotic Regimen on Vancomycin Resistant Enterococcus (VRE) Intestinal Carriage : a Double Blind Randomized Pilot Study
Brief Title: Impact of Probiotic Regimen on Vancomycin Resistant Enterococcus Intestinal Carriage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Olivier LESENS, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHU63-0015
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Vancomycin Resistant Enterococcus Intestinal Carriage
Keywords: Vancomycin Resistant Enterococcus, probiotic

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Lactobacillus casei rhamnosus (strain Lcr 35 LC) — Patients will be blindly randomized to be assigned to a 5 weeks regimen with the probiotic or to a 5 weeks regimen with placebo.

SUMMARY:
This study aims to reduce the duration of VRE intestinal carriage by the administration of Lactobacillus casei rhamnosus (strain Lcr 35 LC). Patients will be blindly randomized to be assigned to a 5 weeks regimen with the probiotic (10 9 lactobacillus bid) or to a 5 weeks regimen with placebo.A stool culture will be performed every week for 5 weeks (during the administration of treatment) then every two weeks until 3 consecutive negative stool culture for VRE.

DETAILED DESCRIPTION:
This study aims to reduce the duration of VRE intestinal carriage by the administration of Lactobacillus casei rhamnosus (strain Lcr 35 LC). Patients will be blindly randomized to be assigned to a 5 weeks regimen with the probiotic (10 9 lactobacillus bid) or to a 5 weeks regimen with placebo.A stool culture will be performed every week for 5 weeks (during the administration of treatment) then every two weeks until 3 consecutive negative stool culture for VRE.

ELIGIBILITY:
Inclusion Criteria:

* Age >18;
* Vancomycin Resistant Enterococcus intestinal carriage

Exclusion Criteria:

* Neutropenia <1000 /mm3,
* Immunosuppressive drugs,
* Inhalation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Reduction of the duration of Vancomycin Resistant Enterococcus intestinal carriage.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier LESENS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Service des Maladies infectieuses et tropicales, Hôpital Gabriel Montpied, Clermont-Ferrand, France

REFERENCES:
- [Derived] Vidal M, Forestier C, Charbonnel N, Henard S, Rabaud C, Lesens O. Probiotics and intestinal colonization by vancomycin-resistant enterococci in mice and humans. J Clin Microbiol. 2010 Jul;48(7):2595-8. doi: 10.1128/JCM.00473-10. Epub 2010 Apr 26. PMID 20421444